CLINICAL TRIAL: NCT06597344
Title: A Phase 3b, Open-label, Single-arm Study in Adolescent and Adult Female Participants to Evaluate Clinical Symptom Improvement and the Safety of Gepotidacin During Treatment of Uncomplicated Urinary Tract Infections (Acute Cystitis)
Brief Title: A Study in Adolescent and Adult Female Participants to Evaluate Clinical Symptom Improvement and the Safety of Gepotidacin During Treatment of Uncomplicated Urinary Tract Infections (Acute Cystitis)
Acronym: SIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 219575
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Urinary Tract Infections
Keywords: Gepotidacin; Uncomplicated Urinary Tract Infection; Acute Cystitis; Symptom Improvement Study (SIS)
MeSH Terms: conditions — Urinary Tract Infections | interventions — gepotidacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gepotidacin (Experimental): Single Arm
  Interventions: Drug: Gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin will be administered.

SUMMARY:
The study will be conducted to evaluate the clinical symptom improvement and safety of oral gepotidacin for treatment of uncomplicated UTI (acute cystitis) in adolescent and adult female participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants having >=12 years of age at the time of signing the informed consent/assent and have a body weight >=40 kilograms (kg).
* The participant has 2 or more of the following clinical signs and symptoms of acute cystitis with onset <96 hours prior to study entry: dysuria, frequency, urgency, or lower abdominal pain.
* The participant has nitrite or pyuria (presence of 3 plus (+)/large leukocyte esterase) on a urine dipstick test from a pre-treatment clean-catch midstream urine sample.
* The participant is capable of giving signed informed consent/assent.
* The participant is female.

Exclusion Criteria:

* The participant resides in a nursing home or dependent care type-facility.
* The participant has a body mass index >=40.0 kilogram per meter square (kg/m^2) or a body mass index >=35.0 kg/m^2 and is experiencing obesity-related health conditions such as uncontrolled high blood pressure or uncontrolled diabetes.
* The participant has a history of sensitivity to the study treatment, or components thereof, or a history of a drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates her participation.
* The participant is immunocompromised or has altered immune defences that may predispose the participant to a higher risk of treatment failure and/or complications.
* The participant has any of the following:
* Poorly controlled asthma or chronic obstructive pulmonary disease; Acute severe pain, Active peptic ulcer disease; Parkinson disease; Myasthenia gravis;
* A history of seizure disorder requiring medications for control (this does not include a history of childhood febrile seizures) Or
* Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention.
* The participant, in the judgment of the investigator, would not be able or willing to comply with the protocol or complete study follow-up.
* The participant has a serious underlying disease that could be imminently life threatening, or the participant is unlikely to survive for the duration of the study period.
* The participant has acute cystitis that is known or suspected to be due to fungal, parasitic, or viral pathogens; or known or suspected to be due to Pseudomonas aeruginosa or Enterobacterales (other than Escherichia coli) as the contributing pathogen.
* The participant has symptoms known or suspected to be caused by another disease process, such as overactive bladder, chronic incontinence, or chronic interstitial cystitis, that may interfere with the clinical efficacy assessments or preclude complete resolution of uUTI symptoms.
* The participant has an anatomical or physiological anomaly that predisposes the participant to UTIs or may be a source of persistent bacterial colonization, including calculi, obstruction or stricture of the urinary tract, primary renal disease (for example [e.g.], polycystic renal disease), or neurogenic bladder, or the participant has a history of anatomical or functional abnormalities of the urinary tract (e.g., chronic vesico-ureteral reflux, detrusor insufficiency).
* The participant has an indwelling catheter, nephrostomy, ureter stent, or other foreign material in the urinary tract.
* The participant who, in the opinion of the investigator, has an otherwise complicated UTI, an active upper UTI (e.g., pyelonephritis, urosepsis), signs and symptom onset >=96 hours before study entry, or a temperature >=101.4 degree Fahrenheit (>=38 Degrees Celsius [°C]), flank pain, chills, or any other manifestations suggestive of upper UTI.
* The participant has known anuria, oliguria, or significant impairment of renal function (creatinine clearance <30 milliliters per minute (mL/min) or clinically significant elevated serum creatinine as determined by the investigator).
* The participant presents with vaginal discharge at Baseline (e.g., suspected sexually transmitted disease).
* The participant has congenital long QT syndrome or known prolongation of the QTc interval.
* The participant has uncompensated heart failure.
* The participant has severe left ventricular hypertrophy.
* The participant has a family history of QT prolongation or sudden death.
* The participant has a recent history of vasovagal syncope or episodes of symptomatic bradycardia or brady arrhythmia within the last 12 months.
* The participant is taking QT-prolonging drugs or drugs known to increase the risk of torsade de pointes (TdP) per the www.crediblemeds.org. "Known Risk of TdP" category at the time of her Baseline Visit, which cannot be safely discontinued from the Baseline Visit to the TOC Visit; or the participant is taking a strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor or a strong P-gp inhibitor
* The participant has a mean triplicate QTc >450 msec or a mean triplicate QTc >480 msec for participants with bundle-branch block.
* The participant has a documented or recent history of uncorrected hypokalemia within the past 3 months.
* The participant has a known ALT value >2 times upper limit of normal (ULN).
* The participant has a known bilirubin value >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* The participant has a current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), including symptomatic viral hepatitis or moderate-to-severe liver insufficiency (Child Pugh class B or C).
* The participant has received treatment with other systemic antimicrobials or systemic antifungals within 1 week before study entry.
* The participant plans to use any of the prohibited medications or nondrug therapies from the Baseline Visit through 7 days after the first dose of study intervention.
* The participant has been previously enrolled in this study or has previously been treated with gepotidacin.
* The participant has participated in a clinical trial and has received an investigational product within 30 days or 5 half-lives, whichever is longer.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 97 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Valencia, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Palm Springs, Florida
  - GSK Investigational Site, Plant City, Florida
  - GSK Investigational Site, Sweetwater, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, West New York, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Forney, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, Mesquite, Texas
  - GSK Investigational Site, Missouri City, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Groups:
- Gepotidacin: Participants with uncomplicated urinary tract infections received 1500 milligram (mg) (2 × 750 mg tablets) Gepotidacin orally as twice daily for 5 days totaling a daily dose of 3000 mg. Each dose was taken after food consumption and with water.
Period: Overall Study
Arm/Group | Gepotidacin
Started | 97
Completed | 96
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gepotidacin
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 45.7 (16.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69
  Black or African American | 20
  Asian | 2
  American Indian or Alaska Native | 1
  Multiple | 1
  Not Reported | 2
  Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Symptom Improvement at 24 Hours (±4 Hours)
Description: Clinical Symptom improvement is defined as a decrease from Baseline in CSS (Clinical Symptom Score) total score of at least 1 point at 24 hours (±4 hours), without the need for other systemic antimicrobials. CSS Score ranges from 0 to 12. Higher scores indicate a higher presence and severity of UTI symptoms.
Time Frame: At 24 hours (h) (±4 h)
Population: Clinically Evaluable (CE) at 24 hours (+4 h) population included all participants in the Intent-to-treat (ITT) population (all participants who enrolled in the study) who adhered to the 2 doses of treatment as prescribed before the 24 hours (±4 hours) CSS assessment (if available), or, before 24 hours (+4 hours) from first dose (if CSS assessment is missing)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gepotidacin
Number analyzed (Participants) | 90
Percentage of participants | 54.4 [43.6 to 65.0]

2. Secondary Outcome: Percentage of Participants Achieving Clinical Symptom Improvement
Description: Clinical Symptom improvement is defined as a decrease from Baseline in CSS total score of at least 1 point at each timepoint(i.e.,48 hours (±4 hours), 72 hours (±4 hours), and 96 hours (±4 hours)), without the need for other systemic antimicrobials. CSS Score ranges from 0 to 12. Higher scores indicate a higher presence and severity of UTI symptoms.
Time Frame: At 48 hours (h) (±4 h), 72 hours (±4 h), 96 hours (±4 h)
Population: CE 48/ 72/ 96 population included all participants in the ITT population who were able to adhere to at least 80% of planned doses of gepotidacin as prescribed before the 48 h (±4 h)/72 h (±4 h)/96 h (+4 h) CSS assessment (if available), or, before 48 h (±4 h)/ 72 h(+4 h)/ 96 h (+4 h) from first dose (if CSS assessment is missing). Only those participants with data available at specified time points have been analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gepotidacin
Number analyzed (Participants) | 90
Percentage of participants
  48 hours (±4 h): number analyzed (Participants) | 89
  48 hours (±4 h) | 79.8 [69.9 to 87.6]
  72 hours (±4 h) | 90.0 [81.9 to 95.3]
  96 hours (±4 h): number analyzed (Participants) | 89
  96 hours (±4 h) | 86.5 [77.6 to 92.8]

3. Secondary Outcome: Percentage of Participants Achieving Clinical Symptom Resolution
Description: Clinical Symptom resolution is defined as a decrease from Baseline to a CSS total score of 0 at each timepoint(i.e., 24 hours (±4 hours), 48 hours (±4 hours), 72 hours (±4 hours), and 96 hours (±4 hours)) without the need for other systemic antimicrobials. CSS Score ranges from 0 to 12. Higher scores indicate a higher presence and severity of UTI symptoms.
Time Frame: At 24 hours (±4 h), 48 hours (±4 h), 72 hours (±4 h), 96 hours (±4 h)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Gepotidacin
Number analyzed (Participants) | 90
Percentage of participants
  24 hours (±4 h) | 3.3 [0.7 to 9.4]
  48 hours (±4 h): number analyzed (Participants) | 89
  48 hours (±4 h) | 12.4 [6.3 to 21.0]
  72 hours (±4 h) | 32.2 [22.8 to 42.9]
  96 hours (±4 h): number analyzed (Participants) | 89
  96 hours (±4 h) | 53.9 [43.0 to 64.6]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious AEs (SAEs) and AE of Special Interest (AESIs)
Description: Adverse Event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose resulted in death,is life-threatening,required hospitalization or prolongation of existing hospitalization,resulted in disability/incapacity,is congenital anomaly/birth defect, other situations which involved medical or scientific judgment or was associated with liver injury and impaired liver function. SAEs are subset of AEs. AEs displayed are TEAEs defined as any AE with an onset date/time on or after treatment start date/time. AESIs include cardiovascular(CV) AEs, gastrointestinal(GI) AEs, clostridioides difficile-associated diarrhea (C. difficile AEs), Acetylcholinesterase Inhibition(AchE-I). AEs were coded using Medical Dictionary for Regulatory Activities (MedDRA). The AE data presented below is of frequency threshold-0%.
Time Frame: Up to 159 days
Population: Safety population included all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin
Number analyzed (Participants) | 97
Participants
  TEAEs | 27
  SAEs | 0
  AESIs | 23

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to 159 days.
Description: Safety population included all enrolled participants who received at least 1 dose of study intervention.
Arm/Group | Gepotidacin
All-Cause Mortality (participants affected / at risk) | 0/97
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 23/97
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin (N=97)
Diarrhoea (Gastrointestinal disorders) | 16 (16)
Flatulence (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT06597344/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT06597344/SAP_001.pdf